CLINICAL TRIAL: NCT03149198
Title: Assessment of the Effectiveness of the Mat Pilates Method in the Treatment of Women With Fibromyalgia in the Santa Cruz City, Rio Grande do Norte, Brazil: A Randomized Controlled Trial
Brief Title: Mat Pilates Method in the Treatment of Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, Prof. Dr., Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE0000
Record Dates: First submitted 2017-04-20; First posted 2017-05-11 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Fibromyalgia, Primary
Keywords: Fibromyalgia, pilates, exercises
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Mat pilates exercises
  Interventions: Other: Mat Pilates exercises
- Control group (Active Comparator): Aquatic aerobic exercises
  Interventions: Other: Aquatic aerobic exercises

INTERVENTIONS:
Other: Mat Pilates exercises — The exercise program based on the pilates method will be performed on the ground in the group room of the FACISA / UFRN Physiotherapy School Clinic in Santa Cruz. The room has ample space and air conditioning for better patient accommodation. The exercises will be performed twice a week for 12 weeks. Each session will last about 50 minutes and will be supervised by a physical therapy student along with the research coordinator. A total of 10 exercises will be performed.
  Arms: Interventional group
Other: Aquatic aerobic exercises — The aerobic exercise program will be held in the therapeutic pool of the Physiotherapy School Clinic of FACISA / UFRN in Santa Cruz. The pool is heated and provides better effects to the proposed treatment.
  The exercises will be performed twice a week for 12 weeks. Each session will last about 50 minutes and will be supervised by another physical therapy student along with the research coordinator.
  Arms: Control group

SUMMARY:
Introduction: Physical exercises have been recommended to improve overall well-being in patients with fibromyalgia, with the main goal of repairing the effects of lack of physical conditioning, and improving symptoms especially pain and fatigue. Very well estimated and widely known are the studies that support the use of the pilates method as effective in improving the symptoms of the disease.

Objective: To evaluate the effectiveness of the soil method in improving pain in women with fibromyalgia in the city of Santa Cruz, RN.

Methodology: This is a randomized controlled trial with blind evaluator, where 60 patients with fibromyalgia diagnosis are divided into two groups. The intervention group, perform an exercise program based on the pilates method in soil and another, considered control group, participate in a program of aerobic exercises in the pool. Both groups conduct supervised exercise programs 2 times a week for a period of 12 weeks. The evaluation instruments used in an EVA (visual pain scale); FIQ Questionnaire - Fibromyalgia Impact Questionnaire; Functional ability by the "Timed Up and Go" test and 6-minute walk test; A quality of sleep by the Pittsburgh Sleep Quality Index (PSQI-BR) and an ESS-BR (Epworth Sleepiness Scale); Finally, a general quality of life for the SF-36.

Statistical analysis: Data are analyzed by t-student, Mann-Whitney test, repeated-measures ANOVA and intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with fibromyalgia diagnosed according to the classification criteria of the American College of Rheumatology,
* aged 18 to 60 years,
* with VAS between 3 and 8,
* who signed the free and informed consent term.

Exclusion Criteria:

* Patients with uncontrolled hypertension;
* Decompensated cardiorespiratory disease;
* History of syncopes or arrhythmias induced by physical exercise;
* Diabetes unbalanced;
* Psychiatric disorders;
* History of regular physical exercise (at least 2 times a week) in the last 6 months
* any other condition that makes it impossible for a patient to perform physical exercises.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 42 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain | baseline
  Visual analogic scale (0-10)
Assessment of Pain | 12 week
  Visual analogic scale (0-10)

SECONDARY OUTCOMES:
Assessment of Function | baseline
  Fibromyalgia Impact Questionnaire
Assessment of Function | 12 Week
  Fibromyalgia Impact Questionnaire
Assessment of Quality of life | baseline
  SF-36 Questionnaire
Assessment of Quality of life | 12 week
  SF-36 Questionnaire
Assessment of Physical Function | baseline
  Timed Up and Go test - This is a performance functional test
Assessment of Physical Function | 12 week
  Timed Up and Go test- This is a performance functional test

CONTACTS AND LOCATIONS:
Locations (1):
- Marcelo Souza, Santa Cruz, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] de Medeiros SA, de Almeida Silva HJ, do Nascimento RM, da Silva Maia JB, de Almeida Lins CA, de Souza MC. Mat Pilates is as effective as aquatic aerobic exercise in treating women with fibromyalgia: a clinical, randomized and blind trial. Adv Rheumatol. 2020 Apr 6;60(1):21. doi: 10.1186/s42358-020-0124-2. PMID 32252822
- [Derived] Silva HJA, Lins CAA, Nobre TTX, de Sousa VPS, Caldas RTJ, de Souza MC. Mat Pilates and aquatic aerobic exercises for women with fibromyalgia: a protocol for a randomised controlled blind study. BMJ Open. 2019 Feb 19;9(2):e022306. doi: 10.1136/bmjopen-2018-022306. PMID 30782866